CLINICAL TRIAL: NCT00960570
Title: An Open-Label Drug Interaction Study to Investigate the Effects of Steady State Fenofibric Acid on the Single-Dose Pharmacokinetics of Efavirenz in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study Between Fenofibric Acid and Efavirenz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-028-08-1018; R08-0056
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: healthy; adult; efavirenz; fenofibric acid; blood levels
MeSH Terms: interventions — efavirenz; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Efavirenz Alone (Active Comparator): Baseline Efavirenz pharmacokinetics.
  Interventions: Drug: Efavirenz 600 mg
- Efavirenz with Steady State Fenofibric Acid (Experimental): Efavirenz pharmacokinetics in the presence of steady state Fenofibric Acid.
  Interventions: Drug: Efavirenz 600 mg; Drug: Fenofibric Acid

INTERVENTIONS:
Drug: Efavirenz 600 mg — Efavirenz 600 mg administered as a single oral dose on the morning of Day 1.
  Arms: Efavirenz Alone
Drug: Efavirenz 600 mg — Co-administered single oral doses of Efavirenz 600 mg and Fenofibric Acid 105 mg on Day 31.
  Arms: Efavirenz with Steady State Fenofibric Acid
Drug: Fenofibric Acid — Co-administered single oral doses of Efavirenz 600 mg and Fenofibric Acid 105 mg on Day 31.
  Arms: Efavirenz with Steady State Fenofibric Acid

SUMMARY:
Efavirenz is predominantly metabolized by cytochrome P450 (CYP) 2B6. Fenofibric Acid is an inhibitor of CYP 2B6. This study will evaluate the effect of multiple doses of fenofibric acid at steady-state on the pharmacokinetics of single-dose efavirenz in healthy adult subjects.

DETAILED DESCRIPTION:
Efavirenz is predominantly metabolized by cytochrome P450 (CYP) 2B6. Fenofibric Acid is an inhibitor of CYP 2B6. This study will evaluate the effect of multiple doses of fenofibric acid at steady-state on the pharmacokinetics of single-dose efavirenz in healthy adult subjects. On study Day 1 after a fast of at least 10 hours, thirty healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one oral dose of efavirenz (1 x 600 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 120 hours post-dose at times sufficient to adequately define the pharmacokinetics of efavirenz. A 21 day washout period will be completed after the first dose of efavirenz on Day 1. On Days 22 through 30, all subjects will receive a single oral dose of fenofibric acid (1 x 105 mg tablet) in the morning without regard to meals. On the morning of Day 31 after a fast of at least 10 hours, all study participants will receive co-administered single oral doses of efavirenz (1 x 600 mg tablet) and fenofibric acid (1 x 105 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 120 hours post-dose at times sufficient to adequately determine the pharmacokinetics of efavirenz. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (seated blood pressure and pulse) will be measured prior to dosing and at approximately 1, 2, 3 and 5 hours post-dose on Days 1 and 31 and prior to dosing and at approximately 1, 2 and 4 hours post-dose on Day 22 to coincide with peak plasma concentrations of both efavirenz and fenofibric acid. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age
* Non-smoking
* Non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures)
* Body mass index (BMI) less than 30
* Medically healthy on the basis of medical history and physical examination
* Hemoglobin > or = to 12g/dL
* Completion of the screening process within 28 days prior to dosing
* Provision of voluntary written informed consent

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to fenofibric acid or efavirenz

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm. D, Principal Investigator — PRACS Insitute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty (30) healthy, non-smoking adult male and female volunteers from the community at-large were enrolled.
Pre-assignment Details: Forty-nine (49) subjects were screened. Nineteen (19) were screen failures.
Groups:
- Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA: On the morning of Day 1, subjects received a single dose of efavirenz 600 mg after an overnight fast of at least 10 hours, followed by a 21 day washout period. On the mornings of Days 22-30, subjects received a dose of fenofibric acid 105 mg without regard to meals. On the morning of Day 31, subjects received a co-administered single oral dose of efavirenz 600 mg and fenofibric acid 105 mg following an overnight fast of at least 10 hours.
Period: Efavirenz Alone
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Started | 30
Completed | 30
Not Completed | 0
Period: 21 Day Washout Period
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Fenofibric Acid Alone
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Started | 28
Completed | 28
Not Completed | 0
Period: 1 Day Period Between Dosing
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Started | 28
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Efavirenz and Fenofibric Acid
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Efavirenz Alone,Fenofibric Acid (FFA) Alone, Efavirenz and FFA
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Efavirenz
Description: The maximum or peak concentration that efavirenz reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing on Days 1 and 31 and then 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, 96 and 120 hours after dose administration.
Population: 30 subjects were enrolled in this study. A total of 6 subjects withdrew. One of those 6 subjects completed all dosing of study interventions but withdrew consent prior to the 8 hour post-dose activities on Day 31.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Efavirenz Alone: On the morning of Day 1, subjects received a single dose of efavirenz 600 mg after an overnight fast of at least 10 hours, followed by a 21 day washout period.
- Efavirenz With Fenofibric Acid: On the morning of Day 31, subjects received a co-administered single oral dose of efavirenz 600 mg and fenofibric acid 105 mg after an overnight fast.
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 24 | 24
ng/mL | 2,461.58 (655.13) | 2,384.79 (573.73)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule for efavirenz.
Time Frame: as for outcome 1
Population: 30 subjects were exposed to study drugs. A total of 6 subjects withdrew. One of those 6 subjects completed all dosing of study medications but withdrew consent prior to the 8 hour post-dose activities on Day 31.
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 24 | 24
ng-hr/mL | 70,144.35 (18,004.09) | 63,313.23 (21,446.35)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. [AUC(0-∞)] was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant for efavirenz.
Time Frame: serial pharmacokinetic blood samples drawn immediately prior to dosing on Days 1 and 31 and then 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 48, 72, 96 and 120 hours after dose administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Efavirenz Alone | Efavirenz With Fenofibric Acid
Number analyzed (Participants) | 24 | 24
ng-hr/mL | 106,689.60 (27,178.11) | 96,382.08 (35,449.72)

ADVERSE EVENTS:
Groups:
- Fenofibric Acid Alone: On the mornings of Days 22-30, subjects received a dose of fenofibric acid 105 mg without regard to meals.
- Efavirenz and Fenofibric Acid: On the morning of Day 31, subjects received a co-administered single oral dose of efavirenz 600 mg and fenofibric acid 105 mg after an overnight fast.
Arm/Group | Efavirenz Alone | Fenofibric Acid Alone | Efavirenz and Fenofibric Acid
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 12 | 7 | 8
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Efavirenz Alone | Fenofibric Acid Alone | Efavirenz and Fenofibric Acid
Tinnitus (Ear and labyrinth disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Diarrhea (Gastrointestinal disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Nausea (Gastrointestinal disorders) | 2/30 (2) | 1/28 (1) | 2/25 (2)
Retching (Gastrointestinal disorders) | 0/30 (0) | 1/28 (1) | 0/25 (0)
Stomach discomfort (Gastrointestinal disorders) | 0/30 (0) | 0/28 (0) | 2/25 (2)
Vomiting (Gastrointestinal disorders) | 0/30 (0) | 2/28 (2) | 1/25 (1)
Chest pain (General disorders) | 0/30 (0) | 1/28 (1) | 0/25 (0)
Feeling cold (General disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Pain (General disorders) | 0/30 (0) | 1/28 (1) | 0/25 (0)
Pyrexia (General disorders) | 0/30 (0) | 1/28 (1) | 1/25 (1)
Sinusitis (Infections and infestations) | 0/30 (0) | 1/28 (1) | 0/25 (0)
Upper respiratory tract infection (General disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Alanine aminotransferase increased (Investigations) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Aspartate aminotransferase increased (Investigations) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Dizziness (Nervous system disorders) | 9/30 (9) | 1/28 (1) | 8/25 (8)
Headache (Nervous system disorders) | 4/30 (4) | 2/28 (2) | 4/25 (4)
Somnolence (Nervous system disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Tremor (Nervous system disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0/30 (0) | 0/28 (0) | 1/25 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/30 (1) | 0/28 (0) | 0/25 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/30 (1) | 1/28 (1) | 1/25 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0/30 (0) | 0/28 (0) | 1/25 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days